CLINICAL TRIAL: NCT06716827
Title: Comparison of Different Teeth Bleaching Methods Performed During Fixed and Clear Aligner Orthodontic Treatments: A Randomized Controlled Clinical Trial
Brief Title: Bleaching Procedures Performed During Treatment With Brackets and Clear Aligners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmet Yağcı (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Sponsor-Investigator, Ahmet Yağcı, PROFESSOR, TC Erciyes University
Organization: TC Erciyes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDK-2023-12793
Record Dates: First submitted 2024-11-26; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Tooth Discoloration
Keywords: Clear aligner treatment; Bleaching; Home bleaching
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional (Experimental): In this group, 14 patients (7 with fixed appliances and 7 with clear aligners) underwent conventional whitening procedures during the treatment process. As the whitening agent, an in-office bleaching system containing 35% hydrogen peroxide (Whiteness HP, FGM) was chosen.
  Interventions: Procedure: In-office bleaching system
- Laser-assisted bleaching (Experimental): In this group, 14 patients (7 with fixed appliances and 7 with clear aligners) underwent laser whitening with a 940 nm diode laser and a 35% hydrogen peroxide gel (Whiteness HP, FGM).
  Interventions: Procedure: Laser-assisted bleaching
- Home bleaching (Experimental): In the home whitening group, 14 patients (7 with fixed appliances and 7 with clear aligners) underwent a 14-day home whitening treatment during the treatment process using a 16% carbamide peroxide gel (Opalescence PF, Ultradent Products Inc., South Jordan, UT, USA).
  Interventions: Procedure: Home-bleaching
- Control (Experimental): The 14 patients randomly selected (7 with fixed appliances and 7 with clear aligners) served as the control group. No whitening procedures were performed on the patients in this group.
  Interventions: Other: Control

INTERVENTIONS:
Procedure: In-office bleaching system — As the whitening agent, an in-office bleaching system containing 35% hydrogen peroxide (Whiteness HP, FGM) was chosen. The gingiva was isolated using an isolation material (Opaldam, Ultradent Products Inc.), which was light-cured with a standard curing light. The whitening gel was applied to the labial surfaces of the maxillary incisors and canines with a 1mm thickness and left for 20 minutes. After cleaning the teeth with an aspiration tip, the whitening procedure was repeated.
  Arms: Conventional
Procedure: Laser-assisted bleaching — Whitening was performed 10 days prior to treatment, with laser treatment applied without removing brackets in the fixed appliance group and without cleaning attachments in the aligner group. The laser was applied to the buccal surface of the teeth with a 1mm distance for 30 seconds in three applications. After a 10-minute rest, the laser procedure was repeated.
  Arms: Laser-assisted bleaching
Procedure: Home-bleaching — The whitening trays were custom-made for the fixed appliance patients, and they used them for 2-4 hours each evening after brushing their teeth. In the transparent aligner group, whitening was done using the aligners worn for treatment.
  Arms: Home bleaching
Other: Control — This group of patients did not undergo any whitening procedures.
  Arms: Control

SUMMARY:
The aim of this study is to compare the effectiveness of different whitening methods used during orthodontic treatment with fixed appliances and clear aligners. It also aims to examine the effect of different whitening methods on white spot lesions and the color change they cause in the teeth.

DETAILED DESCRIPTION:
During orthodontic treatment, if oral hygiene is not properly maintained or in long-term treatments, tooth discoloration may occur. In clear aligner treatment, failure to regularly clean the aligners or the consumption of staining foods and beverages while wearing the aligners can lead to staining and yellowing of the tooth surfaces.

The aim of this study is to compare the effectiveness of different whitening methods used during orthodontic treatment with fixed appliances and clear aligners. It also aims to examine the effect of different whitening methods on white spot lesions using quantitative light-induced fluorescence (QLF) and to evaluate the color changes in the teeth during the treatment process.

ELIGIBILITY:
Inclusion Criteria:

* No previous orthopedic or orthodontic treatment
* Mild or moderate malocclusion
* Non-smokers and non-alcohol consumers
* Consumes no more than 3 cups of tea or coffee per day
* Good oral hygiene and healthy periodontal tissues
* No cavities, restorations, pigmentation, or white spot lesions on the anterior teeth
* Chronological age between 16-30 years, regardless of bone age

Exclusion Criteria:

* Individuals requiring extraction-based treatment
* Individuals who have previously undergone whitening treatment
* Individuals with endogenous tooth discoloration
* Individuals with genetic tooth pigmentation
* Individuals in the mixed dentition phase

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2022-11-09 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
Tooth color measurement | up to 1,5 years
  The screenshots of the scanning records taken at the beginning and end of the treatment were captured, and the L*, a*, b* values were measured using Photoshop software.

SECONDARY OUTCOMES:
QLF(Quantitative light-induced fluorescence) Analysis Score | up to 1 years
  Delta F (ΔF) - The percentage of fluorescence loss relative to a sound tooth

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Faculty of Dentistry, Department of Orthodontics, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Consolaro A, Consolaro RB, Francischone L. Clarifications, guidelines and questions about the dental bleaching "associated" with orthodontic treatment. Dental Press J Orthod. 2013 Sep-Oct;18(5):4-10. doi: 10.1590/s2176-94512013000500002. PMID 24352384
- [Result] Hegedus C, Bistey T, Flora-Nagy E, Keszthelyi G, Jenei A. An atomic force microscopy study on the effect of bleaching agents on enamel surface. J Dent. 1999 Sep;27(7):509-15. doi: 10.1016/s0300-5712(99)00006-8. PMID 10507207
- [Result] Albhaisi Z, Al-Khateeb SN, Abu Alhaija ES. Enamel demineralization during clear aligner orthodontic treatment compared with fixed appliance therapy, evaluated with quantitative light-induced fluorescence: A randomized clinical trial. Am J Orthod Dentofacial Orthop. 2020 May;157(5):594-601. doi: 10.1016/j.ajodo.2020.01.004. PMID 32354432
- [Result] Jadad E, Montoya J, Arana G, Gordillo LA, Palo RM, Loguercio AD. Spectrophotometric evaluation of color alterations with a new dental bleaching product in patients wearing orthodontic appliances. Am J Orthod Dentofacial Orthop. 2011 Jul;140(1):e43-7. doi: 10.1016/j.ajodo.2010.11.021. PMID 21724070